CLINICAL TRIAL: NCT02155751
Title: Bringing an Evidence-based Nutrition and Exercise Lifestyle Intervention Program (NELIP) for Obese Pregnant Women Into Clinical Practice
Brief Title: Bringing NELIP for Obese Pregnant Women Into Clinical Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Debbie Penava, Dr. Debbie Penava, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 102573
Record Dates: First submitted 2013-10-11; First posted 2014-06-04 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Pregnancy
Keywords: Obesity prevention; Nutrition and exercise in pregnancy; Postpartum; Maternal obesity risk
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Full NELIP group (Experimental): These women (n=10) will receive the full NELIP intervention and will be introduced to both the dietary program and the exercise program as described above under "detailed description".
  Interventions: Behavioral: Nutrition Lifestyle Intervention Program (NLIP); Behavioral: Exercise Lifestyle Intervention Program (ELIP)
- Exercise program only/ELIP (Experimental): These women (n=10) will only be given the exercise component (ELIP) of NELIP, as outlined below in interventions. Once dietary intake has been assessed, this group will not be given any dietary intervention but will be encouraged to eat a healthy, balanced diet. Access to the nutritionist in the clinic is available and encouraged.
  Interventions: Behavioral: Exercise Lifestyle Intervention Program (ELIP)
- Nutrition program only/NLIP (Experimental): These women (n=10) will only be given the nutrition program (NLIP) of NELIP as outlined below in intervention. They will be encouraged to be more active but will not be given an exercise intervention.
  Interventions: Behavioral: Nutrition Lifestyle Intervention Program (NLIP)
- Control (No Intervention): A control group (n=30) of obese pregnant women will also be recruited and will be matched by pre-pregnancy BMI, maternal age and parity, with no intervention, but will attend the clinic for standard obstetric care and follow-up.

INTERVENTIONS:
Behavioral: Nutrition Lifestyle Intervention Program (NLIP) — The dietary program will mimic the gestational diabetic meal plan: a) individualize total energy intake with a minimum of 2000 kcal/day (8360 kJ/day), taking into account the usual energy intake as indicated by each dietary assessment (including 3-day food intake records) with a restriction of not more than 33% total energy intake; b) adjust if necessary the total carbohydrate intake to 40-50% of total energy intake, distributing carbohydrate intake throughout the day with three balanced meals, and three snacks per day emphasizing complex carbohydrates and low glycemic index foods; c) adjust the total fat intake to 30% of total energy intake (substituting monounsaturated fatty acids for saturated and trans-fatty acids), with the remaining 30% dedicated to protein intake; and d) meet all micronutrient and fluid needs recommended during pregnancy.
  Arms: Full NELIP group; Nutrition program only/NLIP
Behavioral: Exercise Lifestyle Intervention Program (ELIP) — The exercise program includes a walking program in which pregnant women walk for 25 minutes, 3 to 4 times per week, adding 2 minutes each week, until 40 minutes is reached and then maintained until delivery. Each woman will be given a pedometer and log sheet to keep track of daily steps and to initiate self-monitoring behaviour.
  Arms: Exercise program only/ELIP; Full NELIP group

SUMMARY:
This is a pilot project in which investigators will recruit obese (pre-pregnancy BMI of ≥ 35 kg/m2) women from the newly developed "My Clinic" at London Health Sciences Centre as well as normal obstetrical care at London Health Sciences Centre.

Patients will be randomized to one of three treatment groups: 1) the full Nutrition and Exercise Lifestyle Intervention Program (NELIP), 2) Nutrition program only, or 3) Exercise program only.

The investigators hypothesize that the evidence-based NELIP for obese pregnant women will be feasible to adopt in a clinical setting and will prevent excessive gestational weight gain, gestational diabetes and promote healthy infant growth patterns at the 6 and 12 month milestones. Outcomes may be improved in My Clinic over normal obstetrical care patients with interprofessional services.

DETAILED DESCRIPTION:
Thirty pregnant women (12-16 weeks gestation) with a pre-pregnancy BMI of ≥35 kg/m2 will be recruited from "My Clinic" and normal obstetrical care.

"My Clinic" is a new outpatient obstetrical care clinic being initiated at London Health Sciences Centre for obese women. Women in early pregnancy (12-16 weeks) will be recruited through family physicians' offices from Southwest Ontario to participate in "My Clinic" if their BMI is > or = 35 at the initiation of pregnancy. The clinic will integrate various professional groups currently fractured in their provision of care, including ultrasound, nutrition, social work and obstetrical care to assess and provide care for this group of women, while providing the patients a group atmosphere for regular counselling during their scheduled antenatal visits. The clinic will also offer group counseling sessions for patients covering various topics relating to lifestyle choices including diet and exercise.

Each woman will be screened for medical comorbidities of obesity, including blood pressure measurements and a fasting oral glucose tolerance test to screen for gestational diabetes. Once medically pre-screened with no contraindications to walking regularly, each woman will be approached by a member of the research team. Each woman will record for 3 consecutive days (including one weekend day) a food intake diary and also record the number of steps taken during that same time period, using a pedometer with instructions on how to wear it and record her daily steps. Once these have been returned, the women will be randomized into one of three groups by computer generated model. The order of randomization will be kept in the clinic in opaque envelopes and selected by the research assistant after inclusion in the study is confirmed. The three groups are as described;

1. The NELIP group (N=10) with full intervention (1) will be introduced to a walking program in which they walk for 25 minutes, 3 to 4 times per week, adding 2 minutes each week, until 40 minutes is reached and then maintained until delivery. Each woman will be given a pedometer and log sheet to keep track of daily steps and to initiate self-monitoring behaviour. The dietary program will mimic the gestational diabetic meal plan: a) individualize total energy intake with a minimum of 2000 kcal/day (8360 kilojoule/day), taking into account the usual energy intake as indicated by each dietary assessment (including 3-day food intake records) with a restriction of not more than 33% total energy intake; b) adjust if necessary the total carbohydrate intake to 40-50% of total energy intake, distributing carbohydrate intake throughout the day with three balanced meals, and three snacks per day emphasizing complex carbohydrates and low glycemic index foods; c) adjust the total fat intake to 30% of total energy intake (substituting monounsaturated fatty acids for saturated and trans-fatty acids), with the remaining 30% dedicated to protein intake; and d) meet all micronutrient and fluid needs recommended during pregnancy (2).
2. In order to tease out the effectiveness of the full NELIP, the second group (N=10) will only be given the exercise component (ELIP) of NELIP. Once dietary intake has been assessed, this group will not be given any dietary intervention but will be encouraged to eat a healthy, balanced diet.
3. The third group (N=10) will only be given the nutrition program (NLIP) of NELIP. They will be encouraged to be more active but will not be given an exercise intervention.

A control group (N=30) will also be recruited from the "My Clinic" and other women undergoing care through the obstetrical program at London Health Sciences Centre. The women will be matched by pre-pregnancy BMI, maternal age and parity, with no intervention, but will attend the clinic for standard obstetric care and follow-up.

Women in groups 1-3 will have weekly weight gain recorded until delivery. Infant gender, body weight, length, neonatal morphometrics (birth weight:length ratio, BMI, newborn skinfolds, and circumferences) and placental weight (placenta:birth weight ratio) will be recorded in all women within 6-18 hours of birth. Any interventions or complications at birth will also be recorded. At 6 and 12 months post partum, all maternal-infant pairs (including controls) will be invited to return to the clinic for follow-up. Breast feeding status, maternal weight retention, infant weight/length/BMI/skinfolds/girths and growth patterns will be assessed and compared to the WHO Child Growth Standards for infants based on gender (see above).

All women will complete the Kaiser Physical Activity Questionnaire at entry, 34-36 weeks of gestation and at each follow-up appointment to track changes in physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to "My Clinic" at London Health Sciences Centre
* 18 or older
* 12-20 weeks gestational age
* Pre-pregnancy BMI >= 35kg/m2
* Willing to be randomized

Exclusion Criteria:

* Contraindication to walking regularly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Weight gain in pregnancy | up to 42 weeks
  Average weekly weight gain and total weight gained throughout pregnancy; recorded from initial recruitment (12-20 weeks GA) to date of delivery (up to 42 weeks). This would include approximately 20 weeks on average of follow-up in the clinic, but up to a maximum of 30 weeks total. Women are assessed at 6 months post partum and weight change measured also.

SECONDARY OUTCOMES:
Infant birth weight | Measured at time of birth
  This outcome is measured in grams. Follow-up for infants is also at 6 months of age.
Neonatal morphometrics | Measured at birth, 6 months postpartum, 12 months postpartum
  Includes infant birth weight:length ratio, infant BMI, newborn skinfolds, and circumferences as described prior
Birth complications | Measured at time of birth
Breast feeding | Measured at birth, 6 months postpartum, 12 months postpartum
Maternal weight retention | Measured at 6 and 12 months postpartum
  See above description on weight gain. Analysis will be done and weight gain, retention divided into appropriate groups.
Infant growth | Measured at 6 and 12 months postpartum
  Infant growth will be done in grams and plotted on growth charts, based upon corrected gestational age at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie A Penava, MD, Principal Investigator — London Health Sciences Centre; Michelle Mottola, PhD, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Mottola MF, Giroux I, Gratton R, Hammond JA, Hanley A, Harris S, McManus R, Davenport MH, Sopper MM. Nutrition and exercise prevent excess weight gain in overweight pregnant women. Med Sci Sports Exerc. 2010 Feb;42(2):265-72. doi: 10.1249/MSS.0b013e3181b5419a. PMID 20083959
- [Background] Health Canada. Nutrition for a health pregnancy: National guidelines for the childbearing years. Ottawa (ON): Minister of Public Works & Government Services Canada (CA); 2010.